CLINICAL TRIAL: NCT02269449
Title: RAP and BEAT Clinical Trial (Radial Artery Patency and Bleeding, Effectiveness, Adverse evenT Trial)
Brief Title: Radial Artery Patency and Bleeding, Efficacy, Adverse evenT Trial
Acronym: RAPandBEAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NPO International TRI Network (Network)
Collaborators: European Cardiovascular Research Center (Network); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRI20140920
Record Dates: First submitted 2014-10-07; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Percutaneous Coronary Intervention
Keywords: transradial intervention; radial artery
MeSH Terms: interventions — Hemostasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 6Fr Glidesheath Slender sheath (Experimental): TRI will be performed using a new 6Fr sheath (Glidesheath slender: GSS).
  Interventions: Device: 6Fr Glidesheath Slender sheath
- 5Fr contemporary sheath (Active Comparator): TRI will be performed using a contemporary safety of 5Fr sheath.
  Interventions: Device: 5Fr sheath
- Hemostasis with TR band (Experimental): Hemostasis is achieved by randomization of using TR band (TERUMO) Patent hemostasis.
  Interventions: Procedure: Hemostasis with TR band
- Any hemostasis procedure (Active Comparator): Hemostasis is achieved by randomization of any hemostasis of each hospital's routine procedure.
  Interventions: Procedure: Any hemostasis procedure

INTERVENTIONS:
Device: 6Fr Glidesheath Slender sheath — 6Fr sheath (Glidesheath slender: GSS), which is characterized with the same inner lumen diameter with contemporary 6Fr sheath as well as the sheath outer diameter similar with contemporary 5Fr sheath.
  Arms: 6Fr Glidesheath Slender sheath
Device: 5Fr sheath — 5Fr Hydrophilic coating sheath from Terumo.
  Arms: 5Fr contemporary sheath
Procedure: Hemostasis with TR band — Hemostasis is achieved using TR band (TERUMO) Patent hemostasis.
  Arms: Hemostasis with TR band
Procedure: Any hemostasis procedure — Hemostasis is achieved by any hemostasis of each hospital's routine procedure.
  Arms: Any hemostasis procedure

SUMMARY:
The objectives of this study are to demonstrate the safety and efficacy of the new 6Fr sheath (Glidesheath slender; Terumo, Tokyo,Japan ; GSS) compared with the contemporary 5Fr sheath (Hydrophilic coating sheath from Terumo; Tokyo, Japan (standard of care ; SOC).

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to verbally acknowledge an understanding of the associated risks, benefits and treatment alternatives and he or his legally authorized representative provides written informed consent prior to the randomization, as approved by the appropriate IRB.
* Patient who is expected to diagnose by coronary artery angiography or followed by PCI.
* Patient must agree to undergo all protocol-required follow-up examinations.
* Patient who can accept radial access.

Exclusion Criteria:

* Patient has other medical illness (e.g., cancer or congestive heart failure) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
* Hemodialysis patient
* STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion | Day 1
Local bleeding from puncture site | Day 1

SECONDARY OUTCOMES:
Procedure success rate | Day 1
Vascular access site complication | Day 1
Radial spasm during the index procedure | Day 1
Total Procedure Time | Day 1
Total Amount of Contrast Dye | Day 1
Total Radiation Doses | Day 1
Device failure for the assigned sheath introducer | Day 1
Pain score | Day 1